CLINICAL TRIAL: NCT07191639
Title: Description of the Impact of Symptoms on Quality of Life in HHT Disease: DISQUO
Acronym: DISQUO
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 24-5147
Record Dates: First submitted 2025-08-13; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Hereditary Hemorrhagic Telangiectasia (HHT)
Keywords: Quality of life; HHT
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- HHT patients: completion of the QoL-HHT questionnaire during a consultation at the reference centre
  Interventions: Other: completion of the QOL-HHT questionnaire

INTERVENTIONS:
Other: completion of the QOL-HHT questionnaire — filling in the QOL-HHT questionnaire when they come for consultation

SUMMARY:
In 2017, the ELECT-RO study led, firstly, to the creation of a tool to measure quality of life (QoL) specific to HHT (hereditary haemorrhagic telangiectasia disease), QoL-HHT, based on patients' experiences, their representations and their difficulties. Secondly, the ELECT-RO study demonstrated the validity of the measurement scale, meaning that QoL-HHT does indeed measure patients' QoL and is therefore a reference tool.

QoL-HHT gives investigators a good understanding of the different aspects of patients' QoL (physical limitations, concerns about bleeding, concerns about the evolution of the disease, social relationships, relationships with healthcare professionals and the experience of the disease), whether they are affected or not, at an individual level.

Today, investigators believe it is important to take a more global (population-based) view of the aspects of quality of life affected by HHT. While studies have shown the importance of the role of epistaxis (frequency, duration, intensity, experience) in QoL, what about other symptoms and clinical signs?

The DISQUO study, which the researchers plan to start today, is a follow-up to ELECT-RO. It should enable the researchers to gain a better understanding of the QoL of people with HHT and the impact of each symptom of HHT on patients' QoL.

The DISQUO study will therefore allow the investigators to gain a better understanding of the impact of HHT symptoms on the different areas of patients' QoL.

ELIGIBILITY:
Inclusion Criteria:

* Patient with clinically (presence of at least 3 Curaçao criteria) and/or molecularly confirmed HHT disease
* Patient of legal age (over 18 years old)
* Patient who has received the information and has not objected to taking part in the study

Exclusion Criteria:

* Patients unable to read a questionnaire written in French
* Adults protected by law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Population: Patient with clinically (presence of at least 3 Curaçao criteria) and/or molecularly confirmed HHT disease
  * Patient of legal age (over 18 years old)
  * Patient who has received the information and has not objected to taking part in the study
Sampling Method: Non-Probability Sample
Enrollment: 185 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Description of the quality of life assessed by QOL-HHT scale of HHT patients | Baseline
  the different scores measured by the QOL-HHT scale

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Femme-Mère-Enfant - Centre de référence pour la maladie de Rendu-Osler, Bron, France